CLINICAL TRIAL: NCT03074786
Title: A Phase 2a Crossover Trial Evaluating the Safety of and Adherence to a Vaginal Matrix Ring Containing Dapivirine and Oral Emtricitabine/Tenofovir Disoproxil Fumarate in an Adolescent and Young Adult Female Population
Brief Title: Reversing the Epidemic in Africa With Choices in HIV Prevention (REACH)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was transferred to partner who will conduct under its own IND
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MTN-034/IPM 045
Record Dates: First submitted 2017-02-10; First posted 2017-03-09 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Dapivirine; Contraceptive Devices, Female; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Phase 2a, open-label, multi-site, two-sequence, crossover, randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaginal Matrix Ring (Experimental): Dapivirine vaginal ring containing 25 mg of dapivirine to be replaced each month.
  Interventions: Drug: Dapivirine
- Oral Emtricitanbine/Tenofovir Disoproxil (Experimental): Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) tablets to be taken orally daily
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Dapivirine — Silicone elastomer vaginal matrix ring
  Other Names: Vaginal Ring
  Arms: Vaginal Matrix Ring
Drug: Truvada — Tablets to be taken orally daily
  Other Names: Emtricitabine/tenofovir
  Arms: Oral Emtricitanbine/Tenofovir Disoproxil

SUMMARY:
Participants will be randomized (1:1) to one of two sequences of a vaginal ring (VR) containing 25mg of dapivirine to be inserted monthly for 24 weeks and 200 mg FTC/300 mg TDF oral tablets taken daily for 24 weeks. After completing the randomized sequence of two study product use periods, participants will then select between the two study products to use in the final 24 weeks of the trial. Participants will be able to choose either or neither study product every 4 weeks during the third product use period.

DETAILED DESCRIPTION:
The MTN-034/IPM 045 trial is a multi-site, randomized, two-sequence, three-period, open-label, crossover Phase 2a trial. Young adult (18-21 years old) and adolescent (16-17 years old) female participants will be enrolled in a 2:1 ratio. All the enrolled participants will use both treatment regimens in sequence. All participants will be randomly assigned to one of two treatment regimen sequences to use for the first two study product use periods, and will be able to choose between treatment regimens during the third study product use period. The total length of follow-up is approximately one and a half years which includes up to 72 weeks of product use (two 24-week periods on randomized treatment regimen and one 24-week period on freely chosen treatment regimen) plus an additional week beyond the Period 3 end visit to collect data on any new or worsening AEs.

ELIGIBILITY:
Exclusion Criteria:

1. Become Pregnant and/or use oral PrEP outside the context of study.
2. At Screening or Enrollment, has a positive HIV test.

Inclusion Criteria:

1. Age 16 through 21 years at Enrollment, verified per site standard operation procedures.
2. Able and willing to provide adequate locator information and comply with all study procedural requirements.

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescent and young adult female
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by grade 2 or higher adverse event. | 12 months
  To compare the safety profiles of FTC/TDF oral tablet administered daily and dapivirine vaginal matrix ring (25 mg) inserted for use of each study product in an adolescent and young adult female population

CONTACTS AND LOCATIONS:
Overall Officials: Dianne M Rausch, PHD, Study Director — US National Institutes of Health (NIH)
Locations (1):
- CAPRISA, eThekwini Clinical Research Site, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ngure K, Browne EN, Reddy K, Friedland BA, van der Straten A, Palanee-Phillips T, Nakalega R, Gati B, Kalule HN, Siziba B, Soto-Torres L, Nair G, Garcia M, Celum C, Roberts ST. Correlates of Adherence to Oral and Vaginal Pre-exposure Prophylaxis (PrEP) Among Adolescent Girls and Young Women (AGYW) Participating in the MTN-034/REACH Trial. AIDS Behav. 2024 Sep;28(9):2990-3000. doi: 10.1007/s10461-024-04382-3. Epub 2024 Jun 9. PMID 38852114